CLINICAL TRIAL: NCT02954406
Title: A Phase 1b, Dose Escalation Study to Determine the Recommended Phase 2 Dose of TAK-659 in Combination With Bendamustine (±Rituximab), Gemcitabine, Lenalidomide, or Ibrutinib for the Treatment of Patients With Advanced Non-Hodgkin Lymphoma After At Least 1 Prior Line of Therapy
Brief Title: A Study of TAK-659 in Combination With Bendamustine (+/-Rituximab), Gemcitabine, Lenalidomide, or Ibrutinib for the Treatment of Participants With Advanced Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision, insufficient enrollment, no safety or efficacy concerns.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C34005; U1111-1188-0891 (Other: WHO); 2016-001426-34 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — TAK-659; Bendamustine Hydrochloride; Rituximab; Gemcitabine; Lenalidomide; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 (Experimental): TAK-659 60 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 in a 21-day treatment cycle, for up to 8 cycles. Participants continued to receive TAK-659 monotherapy until they experienced progressive disease (PD) or unacceptable toxicities or up to 39 cycles.
  Interventions: Drug: TAK-659; Drug: Bendamustine
- Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 (Experimental): TAK-659 80 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 in a 21-day treatment cycle, for up to 8 cycles. The TAK-659 was escalated to 80 mg once daily after safety and tolerability of 60 mg dose was determined. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 39 cycles.
  Interventions: Drug: TAK-659; Drug: Bendamustine
- Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 (Experimental): TAK-659 100 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 in a 21-day treatment cycle, for up to 8 cycles. The TAK-659 was escalated to 100 mg once daily after safety and tolerability of 60 mg dose was determined. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 39 cycles.
  Interventions: Drug: TAK-659; Drug: Bendamustine
- Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (Experimental): TAK-659 60 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 along with rituximab 375 mg/m^2, infusion, intravenously, on Day 1 in a 21-day treatment cycle, for up to 8 cycles. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 12 cycles.
  Interventions: Drug: TAK-659; Drug: Bendamustine; Drug: Rituximab
- Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (Experimental): TAK-659 80 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 along with rituximab 375 mg/m^2, infusion, intravenously, on Day 1 in a 21-day treatment cycle, for up to 8 cycles. The TAK-659 was escalated to 80 mg once daily after safety and tolerability of 60 mg dose was determined. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 12 cycles.
  Interventions: Drug: TAK-659; Drug: Bendamustine; Drug: Rituximab
- Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (Experimental): TAK-659 100 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 along with rituximab 375 mg/m^2, infusion, intravenously, on Day 1 in a 21-day treatment cycle, for up to 8 cycles. The TAK-659 was escalated to 100 mg once daily after safety and tolerability of 60 mg dose was determined. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 12 cycles.
  Interventions: Drug: TAK-659; Drug: Bendamustine; Drug: Rituximab
- Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 (Experimental): TAK-659 60 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with gemcitabine 1000 mg/m^2, infusion, intravenously, over 30 minutes on Days 1 and 8 in a 21-day treatment cycle. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 2 cycles.
  Interventions: Drug: TAK-659; Drug: Gemcitabine
- Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg (Experimental): TAK-659 40 mg, immediate-release tablet, orally, once daily on Days 1 to 28 along with lenalidomide 25 mg, capsules orally, once daily on Days 1 to 21 in a 28-day treatment cycle. The TAK-659 60 mg dose was de-escalated to 40 mg in case of dose limiting toxicity or if the starting dose was determined to be not tolerable. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 26 cycles.
  Interventions: Drug: TAK-659; Drug: Lenalidomide
- Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg (Experimental): TAK-659 60 mg, immediate-release tablet, orally, once daily on Days 1 to 28 along with lenalidomide 25 mg, capsules orally, once daily on Days 1 to 21 in a 28-day treatment cycle. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 26 cycles.
  Interventions: Drug: TAK-659; Drug: Lenalidomide
- Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg (Experimental): TAK-659 60 mg, immediate-release tablet, orally, once daily along with ibrutinib 560 mg capsules, orally, once daily on Days 1 to 28 in a 28-day treatment cycle. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 3 cycles.
  Interventions: Drug: TAK-659; Drug: Ibrutinib
- Safety Expansion Phase Cohort B: TAK-659 + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (Experimental): TAK-659 immediate-release tablet, at the MTD/maximally administered dose (MAD)/RP2D determined from Dose Escalation Phase, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 along with rituximab 375 mg/m^2, infusion, intravenously, on Day 1 in a 21-day treatment cycle, for up to 8 cycles in participants (who were to be entered in Phase 2) with advanced FL or MZL. Treatment could then be continued until they experienced PD or unacceptable toxicities or up to 12 cycles in participants who were to be enrolled in the Safety Expansion Phase Cohort.
  Interventions: Drug: TAK-659; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: TAK-659 — TAK-659 immediate release tablet
Drug: Bendamustine — Bendamustine intravenous infusion
  Arms: Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2; Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2; Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2; Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2; Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2; Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2; Safety Expansion Phase Cohort B: TAK-659 + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2
Drug: Rituximab — Rituximab intravenous infusion
  Arms: Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2; Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2; Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2; Safety Expansion Phase Cohort B: TAK-659 + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2
Drug: Gemcitabine — Gemcitabine intravenous infusion
  Arms: Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2
Drug: Lenalidomide — Lenalidomide capsule
  Arms: Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg; Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg
Drug: Ibrutinib — Ibrutinib capsule
  Arms: Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of TAK-659 when administered in combination with bendamustine, bendamustine + rituximab, gemcitabine, lenalidomide, or ibrutinib.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-659. TAK-659 is being tested to treat people who have advanced non-Hodgkin lymphoma. This study will determine the MTD or RP2D for TAK-659 in combination with bendamustine, bendamustine + rituximab, gemcitabine, lenalidomide, and ibrutinib. The study will enroll approximately 96 participants.

Participants will be assigned to one of the 5 combination cohorts:

* Dose Escalation Phase Cohort A: TAK-659 + Bendamustine
* Dose Escalation Phase Cohort B: TAK-659 + Bendamustine + Rituximab
* Dose Escalation Phase Cohort C: TAK-659 + Gemcitabine
* Dose Escalation Phase Cohort D: TAK-659 + Lenalidomide
* Dose Escalation Phase Cohort E: TAK-659 + Ibrutinib This study comprises 2 phases: a dose escalation phase and a safety expansion phase. Participants in all 5 cohorts (Cohorts A-E) will participate in the dose escalation phase of the study. Approximately 12 additional participants with advanced follicular lymphoma (FL) or marginal zone lymphoma (MZL) will be added to Cohort B, in the safety expansion phase.

This multi-center trial will be conducted in North America and Europe. The overall time to participate in this study is approximately 30 months. Participants will make multiple visits to the clinic and will be followed up for safety for 28 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older.
2. In the dose escalation phase, histologically or cytologically confirmed diagnosis of advanced non-Hodgkin lymphoma (NHL) of any histology (with the exception of participants with Waldenström macroglobulinemia [WM] and chronic lymphocytic leukemia [CLL]). In the safety expansion phase for Cohort B, only participants with advanced FL or MZL will be included.
3. Radiographically or clinically measurable disease with at least 1 target lesion per International Working Group (IWG) criteria for malignant lymphoma.
4. In the dose escalation phase, participants who are refractory or relapsed after at least 1 prior line of therapy due to progression, intolerance, or physician/participant decision and for whom no effective standard therapy is available per the investigator's assessment. In the safety expansion phase for Cohort B in participants with FL or MZL, the prior line of therapy is limited to <=1.

   * Either treatment naive to, relapsed/refractory to, or experienced treatment failure due to other reasons with ibrutinib, idelalisib, or any other investigational B-cell receptor (BCR) pathway inhibitors not directly targeting spleen tyrosine kinase (SYK).
   * Pre induction salvage chemotherapy and autologous stem cell transplant (ASCT) should be considered 1 therapy.
   * Any consolidation/maintenance therapy after a chemotherapy regimen (without intervening relapse) should be considered 1 line of therapy with the preceding combination therapy. Maintenance antibody therapy should not be considered a line of therapy.
   * For aggressive NHL (i.e., diffuse large B-cell lymphoma [DLBCL]), single-agent anti-CD20 monoclonal antibody therapy should not be considered a line of therapy. Antibody therapy in participants with indolent NHL (i.e., FL) given as a single agent after disease progression from a prior treatment should be considered a line of therapy.
   * For participants with DLBCL transformed from indolent lymphoma, any treatment received for the indolent disease before the transformation to DLBCL will, in general, not count toward the 2 to 3 prior lines of therapy required for DLBCL in this study.
   * Prior treatment with a regimen that includes the combination drug will not necessarily exclude a participant from that cohort if the investigator views treatment with that agent as appropriate. However, a participant who has a contraindication for a particular combination agent or who has been discontinued from prior therapy with a particular agent for toxicity will not be eligible for inclusion in that particular cohort.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 and life expectancy of greater than 3 months.
6. Participants must have adequate organ function, including the following:

   * Adequate bone marrow reserve: absolute neutrophil count (ANC) greater than or equal to (>=) 1000 per micro liter (/mcL), platelet count >=75,000/mcL (>=50,000/mcL for participants with bone marrow involvement), and hemoglobin >=8 gram per deciliter (g/dL) (red blood cell [RBC] and platelet transfusion allowed >=14 days before assessment).
   * Hepatic: total bilirubin less than or equal to (<=) 1.5×the upper limit of the normal range (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5×ULN.
   * Renal: serum creatinine >=60 milliliter per minute (mL/min) as estimated by the Cockcroft-Gault equation.
   * Others

     * Lipase <=1.5×ULN and amylase <=1.5×ULN with no clinical symptoms suggestive of pancreatitis or cholecystitis.
     * Blood pressure <=Grade 1 (hypertensive participants are permitted if their blood pressure is controlled to <= Grade 1 by hypertensive medications and glycosylated hemoglobin is <=6.5%).
     * Fasting serum glucose level shall be controlled to 130 milligrams per deciliter (mg/dL) during the screening period.
7. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, or
   * Are surgically sterile, or
   * If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

   Male participant, even if surgically sterilized (that is, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
   * Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 international units per liter IU/L or equivalent units of human chorionic gonadotropin [hCG]) at screening.
8. Both men and women in the rituximab combination arm (Cohort B) must practice contraception as described above from the time of signing of the informed consent form (ICF) through 12 months after the last dose of study drug.
9. Female participants should not donate ova from the time of signing the informed consent through 180 days after the last dose of study drug.
10. Male participants should not donate sperm from the time of signing the informed consent through 180 days after the last dose of study drug.
11. Both men and women in the lenalidomide combination arm (Cohort D) must adhere to the guidelines of the RevAssist program (United States participants) or, if not using commercial supplies, must adhere to the Lenalidomide Pregnancy Risk Minimisation Plan as outlined in the Study Manual.
12. Both men and women in the lenalidomide combination arm (Cohort D) must adhere to the guidelines of the RevAssist program (United States participants) or, if not using commercial supplies, must adhere to the Lenalidomide Pregnancy Risk Minimisation Plan as outlined in the Study Manual.
13. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
14. Recovered (that is, <= Grade 1 toxicity) from the reversible effects of prior anticancer therapy.

Exclusion Criteria:

1. Central nervous system (CNS) lymphoma; active brain or leptomeningeal metastases, as indicated by positive cytology from lumbar puncture or computed tomography (CT) scan/magnetic resonance imaging (MRI). Exceptions include those participants who have completed definitive therapy, are not on steroids, have a stable neurologic status for at least 2 weeks after completion of the definitive therapy and steroids, and do not have neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs).
2. Known human immunodeficiency virus (HIV)-related malignancy.
3. Known hypersensitivity (example, anaphylactic and anaphylactoid reactions) to any particular combination drug will result in a participant being ineligible for inclusion in that particular cohort.
4. For participant in the lenalidomide combination arm, demonstrated hypersensitivity (example, angioedema, Stevens-Johnson syndrome, toxic epidermal necrolysis) to lenalidomide.
5. History of drug-induced pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis, organizing pneumonia, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
6. Life-threatening illness unrelated to cancer that could, in the investigator's opinion, make the participant not appropriate for this study.
7. Female participants who are lactating and breast-feeding or a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before the first dose of study drug.
8. Any serious medical or psychiatric illness, including drug or alcohol abuse, that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
9. Known human immunodeficiency virus (HIV) positive.
10. Known hepatitis B surface antigen positive, or known or suspected active hepatitis C infection.
11. Systemic anticancer treatment (including investigational agents) or radiotherapy less than 2 weeks before the first dose of study treatment (<=4 weeks antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T-cell engager agents; <= 8 weeks for cell-based therapy or antitumor vaccine).
12. Prior ASCT within 6 months or prior ASCT at any time without adequate full hematopoietic recovery, defined by the entry criteria in the study, before Cycle 1 Day 1 or allogeneic stem cell transplant any time.
13. Any clinically significant comorbidities, such as uncontrolled pulmonary disease, known impaired cardiac function or clinically significant cardiac disease (specified below), active central nervous system (CNS) disease, active infection, or any other condition that could compromise the participant's participation in the study.
14. Participants with any of the following cardiovascular conditions are excluded:

    * Unstable angina or acute myocardial infarction within 12 months before starting study drug.
    * Current or history of New York Heart Association Class III or IV heart failure.
    * Evidence of current, uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
    * Friderichia corrected QT interval (QTcF) >450 milliseconds (msec) (men) or >475 msec (women) on a 12-lead electrocardiogram (ECG) during the Screening period.
    * Abnormalities on 12-lead ECG including, but not limited to, changes in rhythm and intervals that, in the opinion of the investigator, are considered to be clinically significant.
15. Lack of suitable venous access for the study-required blood sampling for TAK-659.
16. For participants in all combination arms (Cohorts A-E), use or consumption of any of the following substances:

    * Medications or supplements that are known to be inhibitors of P-glycoprotein (P-gp) and/or strong reversible inhibitors of cytochrome P450 (CYP) 3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known) or within 7 days (if a reasonable half-life estimate is unknown) before the first dose of study drug. In general, the use of these agents is not permitted during the study except in cases in which an AE must be managed. See a nonexhaustive list of prohibited strong CYP3A reversible inhibitors and/or P-gp inhibitors based on the US Food and Drug Administration (FDA) Draft Drug-Drug Interactions (DDI) Guidance.
    * Medications or supplements that are known to be strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days or within 5 times the inhibitor or inducer half-life (whichever is longer) before the first dose of study drug. The use of these agents is not permitted during the study. See a list of prohibited strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-glycoprotein (gp) inducers based on the United States (US) Food and Drug Administration (FDA) Draft Drug-drug Interaction (DDI) Guidance.
    * Grapefruit-containing food or beverages within 5 days before the first dose of study drug. Note that grapefruit-containing food and beverages are not permitted during the study.
17. Additionally, for participants in the ibrutinib combination arm (Cohort E), use or consumption of any of the following substances:

    * Medications or supplements that are known to be moderate reversible inhibitors of CYP3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known) or within 7 days (if a reasonable half-life estimate is unknown) before the first dose of study drugs. In general, the use of these agents is not permitted during the study for this combination except in cases in which an adverse event (AE) must be managed. See a list of nonexhaustive moderate CYP3A reversible inhibitors based on the US FDA Draft DDI Guidance.
    * Medications or supplements that are known to be moderate mechanism-based inhibitors or moderate inducers of CYP3A within 7 days or within 5 times the inhibitor or inducer half-life (whichever is longer) before the first dose of study drugs. In general, the use of these agents is not permitted during the study for this combination except in cases in which an AE must be managed. See a list of non-exhaustive moderate CYP3A mechanism-based inhibitors or moderate CYP3A inducers based on the US FDA Draft DDI Guidance.
    * Seville oranges within 5 days before the first dose of study drugs and during the study.
18. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery.
19. Systemic infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
20. Participants with another malignancy within 2 years of study start. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection and are considered disease-free at the time of study entry.
21. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659 including difficulty swallowing tablets or diarrhea >Grade 1 despite supportive therapy.
22. Treatment with high-dose corticosteroids for anticancer purposes within 14 days before the first dose of TAK-659; daily dose equivalent to 10 mg oral prednisone or less is permitted. Corticosteroids for topical use or in nasal spray or inhalers are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (11):
  - University of Arizona Cancer Center, Tucson, Tucson, Arizona
  - University of California San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center (CSMC) - Samuel Oschin Comprehensive Cancer Institute, West Hollywood, California
  - University of Louisville Kentucky James Graham Brown Cancer Center, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - NYU Langone Medical Center - NYU Medical Oncology Associates, New York, New York
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - West Virginia University, Morgantown, West Virginia
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McGill University - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in Canada, Spain, and the United States from 05 March 2017 to 27 July 2020. The study was planned to be conducted in two Phases: Dose Escalation Phase and Safety Expansion Phase, however, per Sponsor's decision, the study was terminated prior to enrollment of participants in the Safety Expansion Phase.
Pre-assignment Details: Participants with a diagnosis of advanced non-Hodgkin lymphoma were enrolled in Dose Escalation Phase Cohorts A, B, C, D and E of study to receive TAK-659 in combination with 1 of 5 combination drugs (bendamustine, bendamustine + rituximab, gemcitabine, lenalidomide, and ibrutinib) to determine the maximum tolerated dose (MTD)/ recommended phase 2 dose (RP2D).
Groups:
- Safety Expansion Phase Cohort B: TAK-659 + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2: TAK-659 immediate-release tablet, at the MTD/maximally administered dose (MAD)/RP2D determined from Dose Escalation Phase, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 along with rituximab 375 mg/m^2, infusion, intravenously, on Day 1 in a 21-day treatment cycle, for up to 8 cycles in participants (who were to be entered in Phase 2) with advanced follicular lymphoma (FL) or marginal zone lymphoma (MZL). Treatment could then be continued until they experienced PD or unacceptable toxicities in participants who were to be enrolled in the Safety Expansion Phase Cohort.
Period: Overall Study
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg | Safety Expansion Phase Cohort B: TAK-659 + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2
Started | 3 | 6 | 6 | 6 | 7 | 3 | 3 | 2 | 4 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 6 | 6 | 7 | 3 | 3 | 2 | 4 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Progressive Disease | 3 | 4 | 3 | 4 | 3 | 3 | 2 | 2 | 1 | 1 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Reason Not Specified | 0 | 0 | 3 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who have received at least 1 dose of study drug.
Groups:
- Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2: TAK-659 60 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 in a 21-day treatment cycle, for up to 8 cycles. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 39 cycles.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7 | 3 | 3 | 2 | 4 | 3 | 43
Age, Continuous [Mean (Full Range); unit: years] | 58.7 [54 to 64] | 61.8 [44 to 76] | 70.5 [57 to 77] | 61.3 [51 to 66] | 57.0 [22 to 72] | 72.7 [63 to 78] | 72.7 [47 to 92] | 58.5 [55 to 62] | 61.0 [47 to 75] | 71.0 [68 to 76] | 64.52 [22 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 2 | 1 | 3 | 0 | 1 | 1 | 15
  Male | 1 | 5 | 3 | 5 | 5 | 2 | 0 | 2 | 3 | 2 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 6 | 6 | 5 | 3 | 3 | 2 | 4 | 3 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  White | 3 | 4 | 6 | 5 | 6 | 3 | 2 | 2 | 4 | 2 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4
  Canada | 3 | 4 | 3 | 5 | 3 | 2 | 0 | 2 | 2 | 2 | 26
  United States | 0 | 2 | 1 | 1 | 3 | 0 | 3 | 0 | 2 | 1 | 13
Height [Mean (Full Range); unit: cm] — Population: Number analyzed is the number of participants with data available for height at the Baseline.
  cm
    number analyzed (Participants) | 2 | 6 | 6 | 6 | 7 | 3 | 3 | 2 | 4 | 3 | 42
    (all) | 171.5 [168 to 175] | 171.7 [155 to 190] | 163.0 [152 to 178] | 170.3 [158 to 176] | 172.7 [164 to 178] | 169.3 [155 to 177] | 154.3 [141 to 165] | 167.5 [167 to 168] | 169.8 [142 to 185] | 164.7 [156 to 174] | 167.5 [141 to 190]
Weight [Mean (Full Range); unit: kg] | 88.0 [58 to 110] | 94.3 [53 to 194] | 76.3 [57 to 108] | 66.7 [49 to 85] | 86.1 [70 to 121] | 87.3 [83 to 94] | 60.0 [49 to 76] | 85.5 [74 to 97] | 90.8 [75 to 119] | 70.0 [50 to 95] | 80.5 [49 to 194]

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Maximum Tolerated Dose (MTD) of TAK-659
Description: MTD was defined as the maximum dose that is determined to be safe and tolerable in different cohorts. Each cohort (A, B, C, D and E) received different escalating doses of TAK-659 in combination with other drugs. For each cohort the maximum tolerated dose of TAK-659 in combination with the other drug/s from the selected dose range is reported.
Time Frame: Cycle 1 (Cohorts A, B and C - each cycle was of 21 days and Cohorts D and E - each cycle was of 28 days)
Population: Dose-limiting toxicity (DLT)-evaluable analysis set: participants who have met the minimum treatment and safety evaluation requirements of the study or who experience a DLT.
Measure: Number; unit: mg
Groups:
- Dose Escalation Phase Cohort A: TAK-659 60-100 mg + Bendamustine 90 mg/m^2: TAK-659 60-100 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 in a 21-day treatment cycle, for up to 8 cycles. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 39 cycles.
- Dose Escalation Phase Cohort B: TAK-659 60-100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2: TAK-659 60-100 mg, immediate-release tablet, orally, once daily on Days 1 to 21 along with bendamustine 90 mg/m^2, infusion, intravenously, over 10 or 60 minutes on Days 1 and 2 along with rituximab 375 mg/m^2, infusion, intravenously, on Day 1 in a 21-day treatment cycle, for up to 8 cycles. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 12 cycles.
- Dose Escalation Phase Cohort D: TAK-659 40-60 mg + Lenalidomide 25 mg: TAK-659 40-60 mg, immediate-release tablet, orally, once daily on Days 1 to 28 along with lenalidomide 25 mg, capsules orally, once daily on Days 1 to 21 in a 28-day treatment cycle. The TAK-659 60 mg dose was de-escalated to 40 mg in case of dose limiting toxicity or if the starting dose was determined to be not tolerable. Participants continued to receive TAK-659 monotherapy until they experienced PD or unacceptable toxicities or up to 26 cycles.
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60-100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60-100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40-60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 15 | 16 | 3 | 6 | 3
mg | NA — Data was not available as MTD was not established. | NA — Data was not available as MTD was not established. | NA — Data was not available as MTD was not established. | NA — Data was not available as MTD was not established. | NA — Data was not available as MTD was not established.

2. Primary Outcome: Dose Escalation Phase: Recommended Phase 2 Dose (RP2D) of TAK-659
Description: The RP2D was the MTD or less. The dose recommended for use in phase 2 studies was analyzed on the basis of the safety, tolerability, and preliminary pharmacokinetic (PK) and efficacy data obtained in phase 1 studies. Each cohort (A, B, C, D and E) received different escalating doses of TAK-659 in combination with other drugs. For each cohort the recommended Phase 2 dose of TAK-659 in combination with the other drug/s from the selected dose range is reported.
Time Frame: Cycle 1 (Cohorts A, B and C - each cycle was of 21 days and Cohorts D and E each cycle was of 28 days)
Population: DLT-evaluable analysis set: participants who have met the minimum treatment and safety evaluation requirements of the study or who experience a DLT.
Measure: Number; unit: mg
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60-100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60-100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40-60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 15 | 16 | 3 | 6 | 3
mg | NA — Data was not available as RP2D was not established. | 60 | NA — Data was not available as RP2D was not established. | NA — Data was not available as RP2D was not established. | NA — Data was not available as RP2D was not established.

3. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-659
Time Frame: Days 1 and 15: Pre-dose and at multiple time points (up to 24 hours) post-dose in Cycle 1 (Cohorts A, B and C - each cycle was of 21 days and Cohorts D and E - each cycle was of 28 days)
Population: Pharmacokinetic (PK) Analysis Set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms(ng)/mL
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7 | 3 | 3 | 1 | 4 | 3
nanograms(ng)/mL
  Cycle 1 Day 1 | 83.61 (92.17) | 89.74 (59.03) | 118.10 (63.83) | 128.58 (27.19) | 142.84 (57.58) | 180.10 (17.93) | 141.27 (296.57) | 139.00 (NA) — The geometric coefficient of variation was not estimable for 1 participant. | 65.03 (80.98) | 120.23 (42.42)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 4 | 5 | 5 | 2 | 2 | 1 | 4 | 2
  Cycle 1 Day 15 | 126.49 (105.13) | 145.03 (96.78) | 187.73 (47.29) | 158.28 (43.71) | 222.96 (31.10) | 223.53 (44.02) | 303.34 (12.39) | 188.00 (NA) — The geometric coefficient of variation was not estimable for 1 participant. | 202.90 (69.27) | 306.59 (66.37)

4. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration for TAK-659
Time Frame: as for outcome 3
Population: PK Analysis Set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7 | 3 | 3 | 1 | 4 | 3
hours (h)
  Cycle 1 Day 1 | 4.00 [4.0 to 4.0] | 2.03 [0.9 to 4.0] | 4.00 [2.1 to 7.7] | 1.10 [0.5 to 4.0] | 2.00 [0.5 to 4.0] | 2.00 [0.1 to 4.0] | 4.13 [0.7 to 4.2] | 0.6 [0.6 to 0.6] | 2.12 [0.7 to 4.0] | 1.00 [0.5 to 2.0]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 4 | 5 | 5 | 2 | 2 | 1 | 4 | 2
  Cycle 1 Day 15 | 4.00 [2.0 to 4.1] | 1.09 [0.3 to 4.5] | 3.83 [0.9 to 7.5] | 1.17 [1.0 to 4.0] | 1.93 [0.8 to 4.0] | 2.47 [0.9 to 4.0] | 2.76 [1.0 to 4.5] | 1.9 [1.9 to 1.9] | 2.08 [0.5 to 8.0] | 1.01 [0.0 to 2.0]

5. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve During Dosing Interval
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×ng/mL
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7 | 3 | 3 | 1 | 4 | 3
h×ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 4 | 5 | 5 | 6 | 3 | 1 | 1 | 4 | 3
  Cycle 1 Day 1 | 1094.51 (52.35) | 1011.49 (53.85) | 1532.34 (65.52) | 852.36 (40.94) | 1455.92 (44.57) | 1444.89 (19.43) | 387.54 (NA) — The geometric coefficient of variation was not estimable for 1 participant. | 1456.03 (NA) — The geometric coefficient of variation was not estimable for 1 participant. | 758.76 (76.63) | 968.82 (36.59)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 4 | 3 | 5 | 5 | 2 | 1 | 1 | 4 | 2
  Cycle 1 Day 15 | 1845.21 (74.17) | 1675.91 (90.89) | 3050.97 (54.46) | 1896.76 (43.15) | 2788.61 (17.61) | 2662.16 (21.31) | 3251.29 (NA) — The geometric coefficient of variation was not estimable for 1 participant. | 2536.48 (NA) — The geometric coefficient of variation was not estimable for 1 participant. | 2578.30 (24.56) | 4218.90 (46.77)

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the response-evaluable population who achieved either complete response (CR), or partial response (PR). CR was defined as the disappearance of all evidence of disease, and PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 123 weeks
Population: Response-evaluable Analysis Set included participants who received at least 1 dose of study drug, had sites of measurable disease at Baseline, and 1 post-baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 3 | 4 | 6 | 5 | 5 | 3 | 2 | 1 | 3 | 2
percentage of participants | 33.3 | 75.0 | 50.0 | 40.0 | 80.0 | 0.0 | 0.0 | 100.0 | 33.3 | 50.0

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documented response to the date of first documented PD. PD was defined as any new lesion or increase by > 50% of previously involved sites from nadir.
Time Frame: Up to 123 weeks
Population: Response-evaluable Analysis Set included participants who received at least 1 dose of study drug, had sites of measurable disease at Baseline, and 1 post-baseline disease assessment. Only responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 1 | 3 | 3 | 2 | 4 | 0 | 0 | 1 | 1 | 1
months | 2.3 [NA to NA] — Due to low number of participants with events upper and lower limits of 95% confidence interval (CI) were not estimable. | 2.8 [1.2 to 4.3] | NA [1.4 to NA] — Median, and upper limits of 95% CI were not estimable as participants were censored. | NA [NA to NA] — Due to low number of participants with events Median, upper and lower limits of 95% CI were not estimable. | 3.9 [2.9 to 4.8] |  |  | 1.8 [NA to NA] — Due to low number of participants with events upper and lower limits of 95% CI were not estimable. | NA [NA to NA] — Due to low number of participants with events median, upper and lower limits of 95% CI were not estimable. | NA [NA to NA] — Median, upper and lower limits of 95% CI were not estimable as participants were censored.

8. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of first drug administration to the date of first documented PD. PD was defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: Up to 123 weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
Number analyzed (Participants) | 3 | 4 | 6 | 5 | 5 | 3 | 2 | 1 | 3 | 2
months | 4.2 [1.3 to 4.7] | 2.7 [2.5 to 5.6] | 9.6 [4.4 to NA] — Due to low number of participants with events the upper limit of 95% CI was not estimable. | 2.6 [1.3 to NA] — Due to low number of participants with events the upper limit of 95% CI was not estimable. | 4.2 [3.8 to 8.3] | 1.3 [0.6 to 1.5] | 1.4 [1.3 to 1.5] | 3.4 [NA to NA] — Due to low number of participants with events upper and lower limits of 95% CI were not estimable. | NA [0.7 to NA] — Due to low number of participants with events the median, and upper limit of 95% CI were not estimable. | 2.7 [NA to NA] — Due to low number of participants with events upper and lower limits of 95% CI were not estimable.

9. Secondary Outcome: Safety Expansion Phase: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of first study drug administration to the date of first documented PD or death due to any cause, whichever occurs first. PD was defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: Up to study completion (Up to 123 weeks)
Population: Data is not available for this outcome measure as the study was terminated prior to start of safety expansion phase.
Arm/Group | Safety Expansion Phase Cohort B: TAK-659 + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form (ICF) through 28 days after the last dose (Up to 123 weeks) of study drug or to the start of subsequent anticancer therapy, whichever occurs first
Description: Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set included participants who have received at least 1 dose of study drug.
Arm/Group | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/6 | 0/6 | 0/6 | 1/7 | 0/3 | 0/3 | 1/2 | 1/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/6 | 4/6 | 2/6 | 6/7 | 2/3 | 1/3 | 1/2 | 0/4 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 6/6 | 7/7 | 3/3 | 3/3 | 2/2 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 (N=3) | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 (N=6) | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 (N=6) | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (N=6) | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (N=7) | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (N=3) | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 (N=3) | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg (N=2) | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg (N=4) | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg (N=3)
Aspergillus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Phase Cohort A: TAK-659 60 mg + Bendamustine 90 mg/m^2 (N=3) | Dose Escalation Phase Cohort A: TAK-659 80 mg + Bendamustine 90 mg/m^2 (N=6) | Dose Escalation Phase Cohort A: TAK-659 100 mg + Bendamustine 90 mg/m^2 (N=6) | Dose Escalation Phase Cohort B: TAK-659 60 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (N=6) | Dose Escalation Phase Cohort B: TAK-659 80 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (N=7) | Dose Escalation Phase Cohort B: TAK-659 100 mg + Bendamustine 90 mg/m^2 + Rituximab 375 mg/m^2 (N=3) | Dose Escalation Phase Cohort C: TAK-659 60 mg + Gemcitabine 1000 mg/m^2 (N=3) | Dose Escalation Phase Cohort D: TAK-659 40 mg + Lenalidomide 25 mg (N=2) | Dose Escalation Phase Cohort D: TAK-659 60 mg + Lenalidomide 25 mg (N=4) | Dose Escalation Phase Cohort E: TAK-659 60 mg + Ibrutinib 560 mg (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 5 | 1 | 2 | 1 | 0 | 2 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 2 | 2 | 3 | 0 | 2 | 0 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 3 | 1 | 0 | 0 | 1 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 4 | 2 | 0 | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 3 | 3 | 5 | 2 | 0 | 0 | 1 | 2
Oedema peripheral (General disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 2 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Swelling face (General disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 6 | 0 | 5 | 0 | 1 | 0 | 1 | 1
Amylase increased (Investigations) | 1 | 2 | 3 | 0 | 3 | 1 | 3 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 3 | 0 | 3 | 0 | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 2 | 3 | 0 | 4 | 0 | 2 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 2 | 4 | 1 | 2 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 5 | 3 | 0 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT02954406/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT02954406/SAP_001.pdf